CLINICAL TRIAL: NCT03627000
Title: Microbiological Epidemiology in Patients Experiencing Microbiological or Clinical Failure Following Reimplantation After a 2-stage Exchange Strategy for Hip or Knee Prosthetic Joint Infection
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Eugénie MABRUT, Clinical Research Assistant, Hospices Civils de Lyon
Other Study IDs: 17-089-2
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Bone and Joint Infection; Bacterial Infections; EPIDEMIOLOGY
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- failure after reimplantation: description of the failure at the reimplantation
  Interventions: Other: failure after reimplantation

INTERVENTIONS:
Other: failure after reimplantation — description of cinical and microbiological failure

SUMMARY:
This study concerns patients having had an infection on their prosthesis (hip, knee,..) and for whom a 2-step exchange of prosthesis has been done.

A 2-step exchange consists in explantation of the prosthesis and implementation of a spacer at the first stage, and reimplantation of a new prosthesis in a second stage. Patients with late prosthetic joint infection are at risk for superinfection at the time of reimplantation.

The aim is to determine the microbiological epidemiology in patients experiencing failure following reimplantation to establish, based on the drug susceptibilities, which cement could be the most active.

ELIGIBILITY:
Inclusion Criteria:

* patients with prosthetic joint infection having had a 2-step exchange at least from the reimplantation, between 2013 and 2015.

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with prosthetic joint infection having had a 2-step exchange managed at the Croix Rousse Hospital from the reimplantation, between 2013 and 2015.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
rate of treatment failure | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption)
  Treatment failure is defined by local clinical and/or microbiological relapse; and/or need for additional surgery; death of septic origin

SECONDARY OUTCOMES:
rate of bacteria involved in microbiological failure | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption)
  description of microbiological failure : bacteria responsible of microbiological failure
rate of clinical failure | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption)
  description of clinical failure

CONTACTS AND LOCATIONS:
Overall Officials: Tristan FERRY, Md,PhD, Principal Investigator — Hospices Civils de Lyon Hôpital de la Croix-Rousse

IPD SHARING:
Plan to Share IPD: Undecided